CLINICAL TRIAL: NCT00081874
Title: Phase I/II Study of RAD001 in Patients With Relapsed or Refractory Acute Myeloid Leukemia, Acute Lymphocytic Leukemia, Chronic Myeloid Leukemia in Blastic-Phase, Agnogenic Myeloid Metaplasia, Chronic Lymphocytic Leukemia, T-Cell Leukemia, or Mantle Cell Lymphoma
Brief Title: RAD001 in Relapsed or Refractory AML, ALL, CML in Blastic-Phase, Agnogenic Myeloid Metaplasia, CLL, T-Cell Leukemia, or Mantle Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0948
Record Dates: First submitted 2004-04-23; First posted 2004-04-27 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2012-10

CONDITIONS: Leukemia; Mantle Cell Lymphoma; Myelofibrosis
Keywords: Leukemia; Mantle cell lymphoma; Myelofibrosis; Relapsed or Refractory Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Chronic Myeloid Leukemia in Blastic-Phase; Agnogenic Myeloid Metaplasia; Chronic Lymphocytic Leukemia; T-Cell Leukemia; RAD001; Everolimus; Afinitor
MeSH Terms: conditions — Leukemia; Lymphoma, Mantle-Cell; Primary Myelofibrosis; Recurrence; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, T-Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental): Phase I: Participants initially treated with 5 mg RAD001 by mouth daily for 28 days.
  Phase II: The MTD (either 5mg or 10mg) administered daily until intolerance or failure or lack of response after 4 cycles of therapy. For assessment purposes, each cycle will comprise a 28-day period.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — Phase I: Starting dose 5 mg by mouth daily for 28 days.
  Phase II: Maximum Tolerated Dose (MTD) from Phase I.
  Other Names: Everolimus; Afinitor

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of RAD001 that can be given as a treatment for leukemia, mantle cell lymphoma, or myelofibrosis. Another goal is to learn how effective the dose that is found is as a treatment.

DETAILED DESCRIPTION:
RAD001 is a new drug that was designed to block proteins that are important in the development and growth of cancer.

If you are eligible to take part in this study, you will receive treatment with RAD001 by mouth every day for as long as you stay on study. Four weeks (28 days) of treatment is considered one course of therapy. The first 3 to 6 participants on study will receive the lowest dose of RAD001. If that dose is safe, the next group of 3 to 6 patients will receive double the dose as the first 3-6 participants. If that dose is safe, all further participants will start treatment at that dose.

While on study, you will have weekly blood tests (about 2 teaspoons). Bone marrow aspirates and/or biopsies, x-rays and/or scans will be performed every 4-12 weeks and as often as the physician feels it is necessary. A physical exam will be done at Weeks 5, 7, 9, 11 and anytime the physician sees fit. Vital signs will be taken every week.

You may be removed from this study if you don't respond after 4 courses of therapy, intolerable side effects occur, or if the disease worsens. Your dose may be temporarily held or decreased if certain side effects occur. If you are benefitting from the therapy, you may continue on it indefinitely as long as continue to benefit.

Once you come off study, a physical exam, measurement of vital signs, a blood test (about 2 teaspoons), a bone marrow aspirate and/or biopsy, x-rays, and/or scans will be done.

This is an investigational study. The FDA has authorized RAD001 for use in research only. A total of 70 -125 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced, relapsed or refractory: acute leukemias (AML, ALL), MDS, CMML in transformation with greater than or equal to 10% peripheral blood/bone marrow blasts, CML in blastic phase, agnogenic myeloid metaplasia (AMM), CLL, T-cell leukemia, or mantle cell lymphoma.
2. Serum bilirubin <= 2 mg/dL, SGOT or SGPT < 3 upper limit of normal, serum creatinine <= 2 mg/dL, unless considered due to organ leukemic involvement or Gilbert's syndrome
3. The effects of RAD001 on the developing human fetus are unknown. For this reason and because inhibitors of mRNA translation are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
4. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had cytotoxic chemotherapy (other than hydroxyurea or corticosteroids) or radiotherapy within 7 days prior to entering the study.
2. Patients may not be receiving any other cytotoxic investigational agents.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to RAD001. RAD001 must not be administered to patients with known hypersensitivity to everolimus, sirolimus or to any of its excipients. Excipients include butylated hydroxytoluene, magnesium stearate, hydroxypropylmethyl-cellulose, crospovidone, and lactose.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Pregnant women are excluded from this study because RAD001 has a potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with RAD001, breastfeeding should be discontinued if the mother is treated with RAD001.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  If either 0 of 3 or 1 of 6 patients assigned to receive dose of 10 mg experiences grade 3 or 4 drug related toxicities, then this dose is the MTD. If greater than 2 patients experience grade 3 or 4 toxicities, either in the first 3 patients or in the first 6 patients, then the MTD is 5 mg.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 28 days
  Number of participants with objective response includes a partial or complete response divided by the total number of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Francis J. Giles, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center's website — http://www.mdanderson.org